CLINICAL TRIAL: NCT03799354
Title: Study on Impact of Maximal Strength Training in Patients With COPD: Physiological and Clinical Implications
Brief Title: Study on Impact of Maximal Strength Training in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICS Maugeri CE 2241
Record Dates: First submitted 2018-12-04; First posted 2019-01-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: rehabilitation; resistive training; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Maximal strenght training (MST) plus endurance training (ET)
  Interventions: Other: Maximal strenght training (MST) plus endurance training (ET)
- Control group (Active Comparator): Endurance training (ET)
  Interventions: Other: Endurance training (ET)

INTERVENTIONS:
Other: Maximal strenght training (MST) plus endurance training (ET) — Patients will perform an addictive out-patients rehabilitative treatment of 8 weeks (3 times/week, ≥20 training sessions) consisting of:
  1. MST- It will consist of four sets of five repetitions on a leg-press with a focus on the rate of force development during the concentric contraction of the quadriceps from a 90° to legs complete extension. The load will be 85-90% of 1RM. When a patient will be able to perform more than five repetitions in a set, the load will be increased. All strength training will be performed on a seated horizontal leg press.
  2. ET - A cycling session will follow the MST and last 40 minutes at constant-load, starting from a load intensity corresponding to patient specific AT. The intensity will be gradually increased with a symptom-based progression.
  Arms: Treatment Group
Other: Endurance training (ET) — Patients will perform a usual out-patients rehabilitative treatment of 8 weeks (3 times/week, ≥20 training sessions). They will perform ET by cycling sessions that will last 40 minutes/each at constant-load, starting from a load intensity corresponding to patient specific AT, assessed during the baseline incremental test. The intensity will be gradually increased during the sessions with a symptom-based progression, according to the protocol by Maltais and coworkers. A 3-min warm-up and cool-down will be provided. Heart rate (HR), blood pressure, oxygen pulsoxymetry, and symptoms by Borg CR10 scale will be monitored at the beginning and end of each session.
  Out of the training-days, both groups will continue their normal daily living with modest regular activity, as recommended by their physician.
  Arms: Control group

SUMMARY:
In the context of pulmonary rehabilitation of COPD patients, recent guidelines and metanalysis describe that Resistance Training (RT) can be successfully performed alone or in conjunction with Endurance Training (ET) without evidence of adverse events.

Maximal Strength Training (MST) is a kind of RT typically performed at ~85-90% of 1RM with maximal velocity to be developed in the concentric phase. Recent literature indicates a significant amelioration on the Rate of Force Development (RFD) after MST in healthy subjects, post-menopausal woman and older populations.

When comparing to the conventional ET, MST generates a little change in muscle mass (no hypertrophy), but a much greater improvement in the RFD. It has been described that neural adjustments play a major role in the MST-induced adaptations. MST is also well documented to improve aerobic endurance by improving walking work efficiency.

Only a small cohort study of COPD patients was conducted, describing that MST can meaningfully improve strength and RFD, with an increase of around 32% for mechanical efficiency and a decrease of the perceived effort during submaximal job. This improvement could determine best performances in daily activities and a best quality of life. The main aims of this physiological pilot randomized controlled trail will be to evaluate feasibility and efficacy of the MST compared to standard ET on strength, effort tolerance, fatigue, economy of walking, dyspnea and risk of falls in a populations of COPD patients, in a short and middle term (6 months).

DETAILED DESCRIPTION:
Exercise intolerance is a cardinal problem existing in patients with Chronic Obstructive Pulmonary Disease (COPD). Moreover, skeletal muscle dysfunction is a common extra-pulmonary manifestation, leading to fatigue, decrease in activity of daily living (ADL) performance and quality of life and increase of risk of falls, mainly in older patients. In the context of pulmonary rehabilitation, recent guidelines and metanalysis describe that Resistance Training (RT) can be successfully performed alone or in conjunction with Endurance Training (ET) without evidence of adverse events.

As concern the RT programs, metanalysis in COPD describe that training have been mainly performed with the lower limbs and the training intensities are heterogeneous, generally ranging from 40% to 70% of 1-Repetition Maximum (1-RM).

Maximal Strength Training (MST) is a RT typically performed at ~85-90% of 1RM with maximal velocity to be developed in the concentric phase. Recent literature indicates a significant amelioration on the Rate of Force Development (RFD) after MST in healthy subjects, post-menopausal woman and older populations.

When comparing to the conventional ET, MST generates a little change in muscle mass (no hypertrophy), but a much greater improvement in the RFD. It has been described that neural adjustments play a major role in the MST-induced adaptations. MST is also well documented to improve aerobic endurance by improving walking work efficiency.

Although the mechanisms at the base of MST effect on the mechanical efficiency have not been completely clarified, there is evidence that changes in the relationships between power and speed bring to a longer relaxation phase inside the cycle of job, improving the recovery between contractions.

In this field, only a small cohort study of COPD patients was conducted describing that MST can meaningfully improve the strength and the RFD, with an increase of around 32% for mechanical efficiency and a decrease of the perceived effort during submaximal job. This improvement could determine best performances in daily activities and a best quality of life. Nevertheless, this study has been conducted only in a small cohort (twelve patients) of patients with COPD and further studies are necessary to define the impact on the different components that determine the effort intolerance.

The main aim of this physiological pilot randomized controlled trail will be to test the feasibility and the efficacy of the MST compared to standard ET on strength, effort tolerance, fatigue, economy of walking, dyspnea and risk of falls in a populations of COPD patients, in a short and middle term (6 months).

ELIGIBILITY:
Inclusion Criteria:

* COPD clinical definition according to GOLD guidelines with forced expiratory volume (FEV1)/ forced vital capacity (FVC) < 70%, and FEV1 < 50% of predicted
* stable clinical condition

Exclusion Criteria:

* pulmonary diseases other than COPD
* type II diabetes or other metabolic diseases
* malign disease
* a respiratory tract infection within the last 4 wks
* long oxygen therapy use.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in walking efficiency | baseline and 8 weeks
  The text will be executed using a portable metabolimeter detecting oxygen consumption (VO2).
  After a 10 min of warm up on a treadmill, the patient will walk 5 min at submaximal steady state walking at 4.5 km/h at 5% incline.
  Using the average of VO2 of the last minute of walking, the walking efficiency will be defined as percentage of change as follows: external work accomplished/ energy expenditure x 100.

SECONDARY OUTCOMES:
Change in Leg Strength by 1-Repetition Maximum on leg press | baseline and 8 weeks
  1-Repetition Maximum (1RM) will be evaluated. 1RM will be measured on a horizontal leg press at a knee angle of 90°. 1RM will be recorded as the heaviest lifted load achieved, applying rest periods of ~4 min between test lifts and increments of 5 kg between each trial until failure.
Change in maximal Rate of Force Development (RFD) | baseline and 8 weeks
  Immediately after the maximal test 1-RM (see above), using the same apparatus, maximal rate of Force Development (RFD) will be assessed using a force platform and applying a load corresponding to 75% of the participant's pre-test 1RM. The subjects will be instructed to execute the lift as rapidly as possible in the concentric phase. RFD will be analyzed as the time difference between 10% and 90% of Peak force.
Change in maximal effort tolerance | baseline and 8 weeks
  It will be evaluated by VO2 consumption on maximal cardiopulmonary exercise test (CPET) on cycloergometer
Change in Constant Load Effort tolerance | baseline and 8 weeks
  It will be evaluated by evaluated by time of execution of Cardiopulmonary Constant-Load Endurance Test
Change in Fatigue (physiological evaluation) | baseline and 8 weeks
  To define peripheral and central component of fatigue, before and after CLET, the investigators will test the difference on force produced during a single twitch superimposed on the Maximal Voluntary Contraction (MVC) and the force produced by the electrically evoked Resting Twitch (RT) produced, at rest, 5 seconds after the MVC.
Change in Fatigue (qualitative evaluation) | baseline and 8 weeks
  Fatigue Severity Scale (scale measuring fatigue, 9-item scale ranging from 7 = absence of fatigue to 63= maximal presence of fatigue)
Change in Muscle volume | baseline and 8 weeks
  Sagittal ultrasound images of the Vastus Lateralis (VL) muscle will be recorded with an 8-12 MHz linear transducer. Images will be obtained with a 90° flexion of hip and knee, at 50% of femur length. The pennation angle (hp) of the VL fascicles will be measured as the angle between the VL muscle fascicles and the deep aponeurosis of the insertion.
Change in Dyspnea | baseline and 8 weeks
  Barthel Index Dyspnea (scale measuring dyspnea during basal ADL, 10-item scale ranging from 0 = absence of dyspnea to 100 = maximal dyspnea)
Concentration of CRP | baseline and 8 weeks
  C reactive protein [CRP] (mg/dl)
Change in Low grade Inflammation | baseline and 8 weeks
  Evaluation of neutrophils/ lymphocytes ratio
Concentration of Tumor necrosis factor alpha | baseline and 8 weeks
  TNF-alpha (pg/ml)
Concentration of Interleukin-6 | baseline and 8 weeks
  IL6 (pg/ml)
Muscular proteolyses by 3-MeH concentration | baseline and 8 weeks
  Evaluation of urinary 3 Methyl-Histine (3-MeH) (micromol/ml)
Change in Balance (qualitative measure) | baseline and 8 weeks
  BERG scale ( scale measuring balance, composed by 14 balance related tasks, ranging from 0 = worse balance to 56= best balance)
Change in quality of life | baseline and 8 weeks
  EuroQol 5-D (scale measuring quality of life, composed by 2 sessions: one of 5 questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with multiple choice ranging from 0 = no problem to 25= very low quality of life and one using Visual Analogic Scale (VAS) to quantify the health status ranging from 0 = worst health condition to 100 = best health condition. The two scale sessions are considered separately.
Patient Satisfaction: Likert Scale | at 8 weeks
  Likert Scale 0-4 ( 0=completely unsatisfied, 4= very satisfied).
Change in Falls | baseline and 8 months
  Evaluation of the rate of falls
Hospitalizations | baseline and 8 months
  Evaluation of the rate of hospitalizations
Mortality | baseline and 8 months
  Evaluation of deaths (number)
Change in Balance (quantitative measure) | baseline and 8 weeks
  The fall risk (FR) assessment will be evaluated by Balance Board.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, MSc, PT, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- ICS Maugeri IRCCS, Respiratory Rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Hoff J, Helgerud J, Wisloff U. Maximal strength training improves work economy in trained female cross-country skiers. Med Sci Sports Exerc. 1999 Jun;31(6):870-7. doi: 10.1097/00005768-199906000-00016. PMID 10378915
- [Background] Hoff J, Tjonna AE, Steinshamn S, Hoydal M, Richardson RS, Helgerud J. Maximal strength training of the legs in COPD: a therapy for mechanical inefficiency. Med Sci Sports Exerc. 2007 Feb;39(2):220-6. doi: 10.1249/01.mss.0000246989.48729.39. PMID 17277584
- [Background] Wang E, Helgerud J, Loe H, Indseth K, Kaehler N, Hoff J. Maximal strength training improves walking performance in peripheral arterial disease patients. Scand J Med Sci Sports. 2010 Oct;20(5):764-70. doi: 10.1111/j.1600-0838.2009.01014.x. PMID 19804581